CLINICAL TRIAL: NCT03421353
Title: A Phase Ib/II, Open-Label, Multicentre Study to Assess Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of AZD9150 Plus Durvalumab Alone or in Combination With Chemotherapy in Patients With Advanced, Solid Tumours and Subsequently in Patients With Non-Small-Cell Lung Cancer
Brief Title: AZD9150 Plus Durvalumab Alone or in Combination With Chemotherapy in Patients With Advanced, Solid Tumours and in Patients With Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5660C00016; REFMAL 558 (Other: Sarah Cannon Development Innovations, LLC); 264476 (Other: Parexel International (IRL) Limited); 2017-004925-34 (EudraCT Number)
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumours
Keywords: AZD9150; Durvalumab; Advanced solid tumours
MeSH Terms: interventions — danvatirsen; durvalumab; Cisplatin; Fluorouracil; Carboplatin; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm A1 (Experimental): Patients will receive AZD9150 every two weeks (Q2W) + durvalumab every four weeks (Q4W). There will be a 1 week AZD9150 lead-in prior to durvalumab dosing.
  Interventions: Drug: AZD9150; Drug: Durvalumab
- Arm A2 (Experimental): Patients will receive AZD9150 once weekly (QW) + durvalumab every three weeks (Q3W) + Cisplatin on Day 1 + 5-flourouracil (5-FU) on Days 1 to 4. This regimen will be repeated every 3 weeks for up to 18 weeks. There will be a 1 week AZD9150 + chemotherapy lead-in prior to durvalumab dosing.
  Interventions: Drug: AZD9150; Drug: Durvalumab; Drug: Cisplatin; Drug: 5-Flourouracil
- Arm A3 (Experimental): Depending on the results of Arm A2, Arm A3 may not be conducted. If Arm A3 is conducted, patients will receive AZD9150 every two weeks (Q2W) + durvalumab every three weeks (Q3W) + cisplatin on Day 1 + 5-flourouracil (5-FU) over Days 1 to 4. This regimen will be repeated every 3 weeks for up to 18 weeks. There will be a 1 week AZD9150 + chemotherapy lead-in prior to durvalumab dosing.
  Interventions: Drug: AZD9150; Drug: Durvalumab; Drug: Cisplatin; Drug: 5-Flourouracil
- Arm A4 (Experimental): Patients will receive AZD9150 every two weeks (Q2W) + durvalumab every three weeks (Q3W) + gemcitabine on Days 1 and 8. This regimen will be repeated every 3 weeks. In addition, the following will be added to the regimen:
  * For cisplatin-eligible patients: cisplatin on Day 1 (every 3 weeks for up to 12-18 weeks); or
  * For cisplatin ineligible patients: carboplatin on Day 1 and Day 8 (every 3 weeks for up to 12-18 weeks)
  There will be a 1 week AZD9150 + chemotherapy lead-in prior to durvalumab dosing.
  Interventions: Drug: AZD9150; Drug: Durvalumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Gemcitabine
- Arm A5 (Experimental): Patients will receive AZD9150 every two weeks (Q2W) plus durvalumab every three weeks (Q3W) plus carboplatin on Day 1 plus nab-paclitaxel on Days 1, 8, and 15 (every 3 weeks for up to 12-18 weeks). There will be a 1 week AZD9150 + chemotherapy lead-in prior to durvalumab dosing.
  Interventions: Drug: AZD9150; Drug: Durvalumab; Drug: Carboplatin; Drug: Nab-paclitaxel
- Arm D: AZD9150 SC (Experimental): Part D will compare the single and steady state pharmacokinetics of AZD9150 given subcutaneously (SC) QW to AZD9150 given by IV QW in combination with durvalumab 1500 mg Q4W. Patients will be randomly assigned to either SC or IV AZD9150.
  Interventions: Drug: AZD9150; Drug: Durvalumab
- Arm D: AZD9150 IV (Experimental): Part D will compare the single and steady state pharmacokinetics of AZD9150 given subcutaneously (SC) QW to AZD9150 given by IV QW in combination with durvalumab 1500 mg Q4W. Patients will be randomly assigned to either SC or IV AZD9150.
  Interventions: Drug: AZD9150; Drug: Durvalumab

INTERVENTIONS:
Drug: AZD9150 — AZD9150 will be administered as a 1-hour intravenous infusion either weekly (QW) or every two weeks (Q2W), depending on which arm the patient is enrolled in.
  AZD9150 will be provided as a liquid drug product in clear glass vials. Each vial will be labelled in accordance with GMP Annex 13 and per country regulatory requirement.
Drug: Durvalumab — Durvalumab will be administered as a 1-hour intravenous infusion either every three weeks (Q3W) or every four weeks (Q4W), depending on which arm the patient is enrolled in.
  Durvalumab will be provided as a solution in clear glass vials. Each vial will be labelled in accordance with GMP Annex 13 and per country regulatory requirement.
  Other Names: MEDI4736
Drug: Cisplatin — Cisplatin will be infused over 30-60 minutes on Day 1.
  Arms: Arm A2; Arm A3; Arm A4
Drug: 5-Flourouracil — 5-flourouracil will be continuously infused over Days 1 to 4 every three weeks for up to 18 weeks.
  Other Names: 5-FU
  Arms: Arm A2; Arm A3
Drug: Carboplatin — Carboplatin will be infused over 30 to 60 minutes on Days 1, 8, and 15, depending on which arm the patient is enrolled in, for up to 18 weeks.
  Arms: Arm A4; Arm A5
Drug: Gemcitabine — Gemcitabine will be infused over 30 minutes on Days 1 and 8 for up to 18 weeks.
  Arms: Arm A4
Drug: Nab-paclitaxel — Nab-paclitaxel will be infused over 30 to 40 minutes on Days 1, 8, and 15 for up to 18 weeks.
  Arms: Arm A5

SUMMARY:
This is a phase Ib/II, open-label multicentre study to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumour activity of AZD9150 plus durvalumab alone or in combination with chemotherapy in patients with advanced, solid tumours and subsequently in patients with non-small-cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This international, multicenter study was originally intended to be conducted in four parts, designated as Parts A, B, C, and D. The protocol was amended in December 2018 to remove Parts B and C. Parts B and C were intended to evaluate patients with locally advanced or metastatic Stage IV NSCLC; however, these parts of the study will not be conducted.

Part A of this study will evaluate the safety and tolerability of durvalumab and AZD9150 with and without selected chemotherapy regimens, and will include patients with advanced solid malignancies that are refractory to standard therapy or for whom no standard of care (SOC) regimen currently exists.

Part D will compare the relative bioavailability of the AZD9150 subcutaneous (SC) versus intravenous (IV) formulations in patients with confirmed solid malignancies that are refractory to standard therapy or for whom no SOC regimen currently exists. Approximately 50 to 62 PK-evaluable patients will be enrolled in Part D. Patients will be randomly assigned to either SC or IV AZD9150. For Part D, the PK Analysis set will include all patients who receive both study drugs (both AZD9150 and durvalumab) and have at least one PK sample collection.

A complementary anti-tumour strategy will be used in this study with 2 immuno-therapeutics applied to restore effective anti-tumour immunity at 2 distinct stages: promoting the effector function of T-cell responses with an anti-PD-L1 mAb, durvalumab, while hindering immune escape in the tumour bed with AZD9150. In addition, chemotherapy will be added to this combination to investigate possible future enhancement of response. In preclinical models, conventional platinum-based chemotherapy has been shown to induce T-cell activation through the release of tumour-specific antigens during cancer cell death. The elimination of persistent tolerogenic tumour antigen environment via chemotherapy-induced debulking may also play a role in generating an effective immune response. In this setting, immunotherapy has the potential to mount an ongoing and dynamic immune response that can kill tumour cells for an extended time.

Part A of the study will be conducted in five arms, designated Arms A1, A2, A3, A4, and A5. The primary objective of Part A is to assess the safety and tolerability, and determining the maximum tolerated dose/recommended phase 2 dose (MTD/RP2D) of AZD9150 plus durvalumab in patients with advanced solid malignancies. In addition, another primary objective is to assess the safety and tolerability, and determine the maximum tolerated dose/recommended phase 2 dose (MTD/RP2D) of AZD9150 plus durvalumab in combination with standard chemotherapy regimens in patients with advanced solid malignancies. Approximately 30 to 78 DLT-evaluable patients will be enrolled in Part A.

In Arm A1, patients will receive AZD9150 by (IV) infusion Q2W + durvalumab by IV infusion Q4W. Chemotherapy will not be given in Arm A1.

Arm A2 patients will receive AZD9150 IV QW + durvalumab IV Q3W, cisplatin by slow IV infusion over 1-4 hours on Day 1 + 5-fluorouracil (5FU) by continuous IV infusion over 96 hours (Days 1 through 4, repeated every 3 weeks for up to 18 weeks). In Arm A2 there will be a AZD9150 + chemotherapy lead-in period prior to durvalumab dosing. The last chemotherapy dose will be given in Week 15. After discontinuation of chemotherapy the regimen will include AZD9150 IV QW + durvalumab IV Q4W. Administration of durvalumab will continue Q3W through Week 19, at which time the schedule will switch to Q4W (e.g., Week 23, 27, 31, etc.).

Depending on the results from Arm A2, Arm A3 may not be conducted. If the Safety Review Committee (SRC) decides to open Arm A3, the SRC will determine the starting dose. Patients will be administered one of the following 4 chemotherapy regimens in combination with AZD9150 and durvalumab appropriate for their tumour type:

* In Arm A3, patients will receive cisplatin by slow IV infusion over 1-4 hours on Day 1 + 5FU by continuous IV infusion over 96 hours (Days 1 through 4, repeated every 3 weeks for up to 18 weeks).
* In Arm A4, patients will receive gemcitabine by IV infusion over 30 minutes on Days 1 and 8 every 3 weeks for 12 to 18 weeks, plus either:

  * for cisplatin-eligible patients: cisplatin IV over 30 minutes on Day 1 (every 3 weeks for up to 12 to 18 weeks); or
  * for cisplatin-ineligible patients: carboplatin IV over 30 to 60 minutes on Day 1 (every 3 weeks for up to 12 to 18 weeks).
* In Arm A5, patients will receive carboplatin at AUC 5 IV over 30 to 60 minutes on Day 1 + nab-paclitaxel IV over 30 to 40 minutes on Days 1, 8, and 15 (every 3 weeks for up to 12 to 18 weeks)

There will be an AZD9150 7-day lead-in period (termed Week 0) in all arms in all parts of the study. AZD9150 will be given IV on Days 1,3, and 5 of the lead-in week. When chemotherapy is administered, the dosing of chemotherapy will also commence during the lead-in period with AZD9150. In Arm A2 of Part A, dosing with AZD9150 IV, durvalumab, and chemotherapy will commence on Day 1 of Week 0. In Part D, dosing with AZD9150 IV or SC will commence on Day 1 of Week 0

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible to be included in the study only if all of the following inclusion criteria and none of the exclusion criteria apply.

1. Signed and dated informed consent. For inclusion in the optional pharmacogenetic research, patients must provide informed consent for the genetic sampling and analyses.
2. ≥ 18 years of age.
3. An Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Minimum life expectancy of 12 weeks
5. Part A of the study will include patients that have histological confirmation of a solid malignancy [other than Hepatocellular Carcinoma (HCC)] that is refractory to standard therapy or for which no standard of care regimen currently exists.
6. Part D of the study will include patients with histological confirmation of a solid malignancy (other than HCC) that are refractory to standard therapy of for which no standard of care regimen currently exists.
7. Willing to undergo mandatory biopsy at screening and on treatment. Part A only: the first 3 subjects in each arm are exempt from this requirement. Patients in Part D are exempt from this biopsy requirement.
8. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes that must have short axis ≥15 mm) with computerised tomography (CT) or magnetic resonance imaging (MRI) that is suitable for accurate repeated measurements.
9. Females should be using adequate contraceptive measures, should not be breast feeding, and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinising hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.
10. Male patients must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign consent) and for 20 weeks after the last dose of study treatments.

Exclusion Criteria

Patients should not enter the study if any of the following exclusion criteria are fulfilled.

1. Involvement in the planning and/or conduct of the study (applies to AstraZeneca and/or Sarah Cannon Development Innovations staff and/or staff at the study site).
2. Previous enrolment in the present study.
3. Herbal preparations are not allowed throughout the study. These herbal medications include but are not limited to St. John's wort, kava, ephedra (mahung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto and ginseng. Patients should stop using herbal medications 7 days prior to the first dose of study treatment.
4. Brain metastases or spinal cord compression unless asymptomatic and not requiring steroids for at least 14 days prior to start of study treatment.
5. With the exception of alopecia and haemoglobin (Hb) ≥ 9 mg/dL and < 10 mg/dL, any unresolved toxicities from prior therapy CTCAE Grade > 1 at the time of starting study treatment.
6. Active interstitial lung disease (ILD)/pneumonitis or a prior history of ILD/pneumonitis requiring treatment with steroids.
7. Patients receiving any concurrent chemotherapy, radiotherapy, immunotherapy, or biologic, or hormonal therapy for cancer.

   * Concurrent use of hormones for noncancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable. The dose of systemic corticosteroids must not exceed 10 mg of prednisone equivalent.
   * Patients in Part A and Part D with radically-treated prostate cancer may continue androgen deprivation therapy (ADT).
8. Patients must have completed any previous cancer-related treatments before enrolment. The following intervals between the end of the prior treatment and first dose of study drug must be observed:

   * Port-a-cath placement: no waiting is required
   * Minor surgical procedures (as defined by the Medical Monitor): 7 postoperative days
   * Major surgery (as defined by the Medical Monitor): ≥4 weeks
   * Radiotherapy: ≥4 weeks (patients who receive palliative radiation for nontarget tumour lesions need not be subjected to this washout period and can be enrolled immediately)
   * Chemotherapy: ≥ 21 days or 5 half-lives (whichever is longer) from the first dose of study drug
   * Immunotherapy and/or anticancer therapy with agents including mAbs ≥4 weeks
   * Current or prior use of immunosuppressive medication within 14 days before first dose of durvalumab The following are exceptions to this criterion:

     * Use of intranasal, inhaled, topical corticosteroids, local steroid injections (e.g., intra articular injections)
     * Systemic corticosteroids at physiologic doses below 10 mg/day of prednisone or equivalent is permitted
     * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) are permitted
9. For Part A and Part D patients who have received more than 3 prior cytoreductive chemotherapy regimens.
10. Has active or prior documented autoimmune disease within the past 2 years with the exceptions of vitiligo, Graves' Disease, and/or psoriasis not requiring systemic treatment
11. Has active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
12. Has a history of primary immunodeficiency
13. Has undergone an organ transplant that requires use of immunosuppressive treatment
14. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) calculated using Fridericia's formula (QTcF) of >450 msec for males and >470 msec for females obtained from 3 electrocardiograms (ECGs) taken over 5 minutes
    * Any clinically important abnormalities in rhythm, conduction or morphology of a resting ECG, e.g., complete left bundle branch block, third degree heart block, that in the opinion of the Investigator renders the patient unsuitable for participation in the study
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age
    * Any concomitant medication with known or possible risk of prolonging the QT interval.
15. Inadequate organ and marrow function as demonstrated by any of the following laboratory values. Transfusions intended to elevate any parameters below solely for the intent of meeting study eligibility are not permitted.

    * Leukocytes <3.0 x 10(exp 9)/L
    * Absolute neutrophil count <1.5 x 10(exp 9)/L
    * Platelet count <100 x 10(exp 9)/L
    * Haemoglobin <90 g/L
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
    * Total bilirubin >1.5 times ULN if no liver metastases or 3 times ULN in the presence of liver metastases or documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia)
    * Creatinine outside normal limits OR, if creatinine outside normal limits, a creatinine clearance <60 mL/min (measured by 24-hour urine collection or calculated by Cockcroft and Gault equation (Cockcroft and Gault 1976).
16. Has a history of allergic reactions attributed to the study treatments (AZD9150 or durvalumab), assigned chemotherapy agents, their compounds, or agents of similar chemical or biologic composition (e.g., antibody therapeutics)
17. Suffers from a comorbidity that in the opinion of the Investigator or Medical Monitor renders the patient unsuitable for participation in the study. Such comorbidity may include, but is not limited to, uncontrolled intercurrent illness such as active infection, severe active peptic ulcer disease or gastritis, myocardial infarction within 6 months before entry, congestive heart failure, symptomatic congestive heart failure, active cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
18. As judged by the Investigator, has any evidence of severe or uncontrolled diseases, or has an active viral infection of human immunodeficiency virus (HIV), human papilloma virus (HPV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV)].
19. Active infection including tuberculosis (clinical evaluation that included clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice).
20. Has received a live attenuated vaccine within 28 days before the first dose of study drug
21. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Tolerated Dose (MTD) in subjects receiving AZD9150 plus durvalumab and AZD9150 plus durvalumab plus chemotherapy. | Through study completion (an average of 6 months). Dose-limiting toxicities (DLTs) will be assessed through 5 weeks for patients who do not receive chemotherapy or 3 weeks for patients receiving chemotherapy.
  The Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) will be determined by assessment of the incidence of dose-limiting toxicities (DLTs). DLTs may come from the incidence and severity of adverse events (AEs) and serious adverse events (SAEs), the change from baseline in vital signs, clinical chemistry, haemotology, and urinalysis parameters will be evaluated for each treatment arm in Part A of the study.
Part D: Area under the plasma concentration versus time curve at steady state [AUC(ss)] of AZD9150 administered once per week in combination with durvalumab. | Blood samples for the PK analysis of AZD9150 will be collected at prespecified intervals during Weeks 0, 1, 5, 6, and 9.
  Pharmacokinetic parameters will be derived from the measured plasma concentration of AZD9150. The area under the plasma concentration versus time curve [AUC(ss)] will be compared in subjects receiving AZD9150 subcutaneoulsy vs. intravenously.
Part D: Minimum plasma concentration at steady state [Ctrough (ss)] of AZD9150 administered once per week in combination with durvalumab. | Blood samples for the PK analysis of AZD9150 will be collected at prespecified intervals during Weeks 0, 1, 5, 6, and 9.
  Pharmacokinetic parameters will be derived from the measured plasma concentration of AZD9150. The minimum plasma concentration of AZD9150 at steady state [Ctrough(ss)] will be determined for subjects receiving AZD9150 once per week in combination with durvalumab.

SECONDARY OUTCOMES:
Part A: Disease Control Rate (DCR) | 12 weeks
  Efficacy parameters as defined by RECIST v1.1 for each combination (with and without chemotherapy) and schedule include: disease control rate (DCR) at 12 weeks, duration of overall response (DOR), and progression-free survival (PFS).
Part A: Duration of Overall Response (DoR) | Throughout the study (approximately 6 months).
  Efficacy parameters as defined by RECIST v1.1 for each combination (with and without chemotherapy) and schedule include: disease control rate (DCR) at 12 weeks, duration of overall response (DOR), and progression-free survival (PFS).
Part A: Progression-Free Survival (PFS) | From the date of documented complete response or partial response, whichever comes first, until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Efficacy parameters as defined by RECIST v1.1 for each combination (with and without chemotherapy) and schedule include: disease control rate (DCR) at 12 weeks, duration of overall response (DOR), and progression-free survival (PFS).
Part A: AZD9150 anti-drug antibody titres | Blood samples for AZD9150 anti-drug antibodies (ADAs) will be collected predose on prespecified dosing days up to 9 weeks.
  Unwanted immunogenicity in the form of anti-drug-antibodies (ADAs) will be assessed.
Part A: Durvalumab anti-drug antibody titres | Blood samples for durvalumab anti-drug antibodies (ADAs) will be collected predose on prespecified dosing days up to 13 weeks.
  Unwanted immunogenicity in the form of anti-drug-antibodies (ADAs) will be assessed.
Part A: Baseline tumour PD-L1 expression | Pre-dose
  Baseline tumour PDL1 expression will be evaluated for potential correlation with drug activity or the ability to prospectively identify patients likely to respond to treatment.
  Immunohistochemistry (IHC) for PD-L1 will be carried out using a tumour sample from an archival biopsy or one taken at screening.
Part A: STAT3 protein in tumour biopsies | Predose and 3 weeks after start of treatment
  STAT3 knockdown will be assessed in tumour biopsies taken on-treatment at Week 3, Day 1. Baseline and on-treatment biopsies will be used to measure STAT3 expression levels by immunohistochemistry.
Part A: Peak plasma concentration (Cmax) of AZD9150 after single-dose. | Blood samples for the PK analysis of AZD9150 will be collected at prespecified intervals during Weeks 0, 1, 5, 6, and 9.
  The peak plasma concentration (Cmax) of AZD9150 after single dose and at steady state after multiple doses in combination with durvalumab Q4W will be determined.
Part A: Trough plasma concentration (Ctrough) of AZD9150 after single-dose. | Blood samples for the PK analysis of AZD9150 will be collected at prespecified intervals during Weeks 0, 1, 5, 6, and 9.
  The trough plasma concentration (Ctrough) of AZD9150 after single dose and at steady state after multiple doses in combination with durvalumab Q4W will be determined.
Part A: Peak plasma concentration (Cmax,ss) of AZD9150 after multiple doses. | Blood samples for the PK analysis of AZD9150 will be collected at prespecified intervals during Weeks 0, 1, 5, 6, and 9.
  The peak plasma concentration (Cmax,ss) of AZD9150 at steady state after multiple doses in combination with durvalumab Q4W will be determined.
Part A: Trough plasma concentration (Ctrough,ss) of AZD9150 after multiple doses. | Blood samples for the PK analysis of AZD9150 will be collected at prespecified intervals during Weeks 0, 1, 5, 6, and 9.
  The trough plasma concentration (Ctrough,ss) of AZD9150 at steady state after multiple doses in combination with durvalumab Q4W will be determined.
Part A: Area under the plasma concentration versus time curve (AUC) of AZD9150 after single-dose. | Through study completion (an average of 6 months)
  The area under the plasma concentration versus time curve (AUC) of AZD9150 after single-dose given in combination with durvalumab Q4W will be determined.
Part A: Area under the plasma concentration versus time curve [AUC(ss)] at steady state after multiple doses. | Through study completion (an average of 6 months)
  The area under the plasma concentration versus time curve [AUC(ss)] of AZD9150 at steady state after multiple in combination with durvalumab Q4W will be determined.
Part D: Injection site tolerability for patients receiving subcutaneous injections. | Through study completion (an average of 6 months)
  Pain, tenderness, redness, and other symptoms will be assessed for subcutaneous injection of AZD9150.
Part D: The incidence of adverse events (AEs) in subjects receiving AZD9150. | Through study completion (an average of 6 months)
  The incidence of adverse events will be determined for each treatment arm in Part D of the study.
Part D: The incidence of serious adverse events (SAEs) in subjects receiving AZD9150. | Through study completion (an average of 6 months)
  The incidence of serious adverse events will be determined for each treatment arm in Part D of the study.
Part D: Peak plasma concentration (Cmax) of AZD9150 after single-dose. | Through study completion (an average of 6 months)
  The peak plasma concentration (Cmax) of AZD9150 after single dose and at steady state after multiple doses when given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: Peak plasma concentration (Cmax,ss) of AZD9150 at steady state after multiple doses. | Through study completion (an average of 6 months)
  The peak plasma concentration (Cmax) of AZD9150 after single dose and at steady state after multiple doses when given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: Time to peak plasma concentration (tmax) of AZD9150 after single-dose. | Through study completion (an average of 6 months)
  The time to peak plasma concentration (tmax) of AZD9150 after single dose when given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: Area under the plasma concentration versus time curve [AUC(0-inf)] after single-dose. | Through study completion (an average of 6 months)
  The area under the plasma concentration versus time curve from zero time to infinity [AUC(0-inf)] of AZD9150 after single dose given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: Area under the plasma concentration versus time curve [AUC(ss)] at steady state after multiple doses. | Through study completion (an average of 6 months)
  The area under the plasma concentration versus time curve [AUC(ss)] of AZD9150 at steady state after multiple doses given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: Area under the plasma concentration versus time curve [AUC(0-t)] after single-dose. | Through study completion (an average of 6 months)
  The area under the plasma concentration versus time curve from zero time to time t [AUC(0-t)] of AZD9150 after single dose given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: Area under the plasma concentration versus time curve from time zero to 48 hours [AUC(0-48] after single-dose. | Through study completion (an average of 6 months)
  The area under the plasma concentration versus time curve from zero time to 48 hours [AUC(0-48)] of AZD9150 after single dose given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: The systemic clearance (CL) of AZD9150 after single-dose. | Through study completion (an average of 6 months)
  The systemic clearance (CL) after single-dose will be calculated for AZD9150 given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: The systemic clearance [CL(ss)] of AZD9150 after multiple doses. | Through study completion (an average of 6 months)
  The systemic clearance [CL(ss)] after multiple doses will be calculated for AZD9150 given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: The apparent systemic clearance (CL/F) of AZD9150 after single-dose. | Through study completion (an average of 6 months)
  The apparent systemic clearance (CL/F) after single-dose will be calculated for AZD9150 given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: The volume of distribution (Vz/F) of AZD9150 after single-dose. | Through study completion (an average of 6 months)
  The volume of distribution (Vz/F) after single-dose will be calculated for AZD9150 given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: The mean residence time (MRT) of AZD9150 after single-dose. | Through study completion (an average of 6 months)
  The mean residence time (MRT) after single-dose will be calculated for AZD9150 given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: The elimination half-life (t1/2) of AZD9150 after single-dose | Through study completion (an average of 6 months)
  The elimination half-life (t1/2) after single-dose will be calculated for AZD9150 given subcutaneously QW relative to intravenous administration QW in combination with durvalumab Q4W will be determined.
Part D: Injection site tolerability of AZD9150 given by subcutaneous injection every 4 weeks relative to AZD9150 200 mg IV QW in | Through study completion (an average of 6 months)
  Injection site tolerability will be assessed by careful visual observation of both subcutaneous and intravenous injection sites and questioning the patient about adverse events at the injection site.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Johnson, M.D., Principal Investigator — Tennessee Oncology
Locations (6):
- United States (6):
  - Research Site, Lafayette, Indiana
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: CSR_synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5660C00016&attachmentIdentifier=b344a4df-559e-4edc-bad5-98b8d23133dc&fileName=D5660C00016_CSR_synopsis_Redaction_Jan2022_Redacted.pdf&versionIdentifier=